CLINICAL TRIAL: NCT06461065
Title: Evaluation of Neurodevelopmental Trajectories in Children According to the Glycemic Profile Associated With Different Early Treatment Modalities in Children With Type 1 Diabetes (T1DM)
Acronym: PROCEDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation Francophone pour la Recherche sur le Diabete (Other); mylife Diabetes Care AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APHP230422
Record Dates: First submitted 2024-05-31; First posted 2024-06-14 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Diabetes
Keywords: Diabetes; Children; insulin therapy; cognitive development
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AIDS group (Experimental): patients with T1DM with automatized insulin delivery systems (AIDS)
  Interventions: Device: AIDS; Other: Brain MRI
- TS group (Other): patients with T1D treated with insulin pumps + blood glucose sensors with the option of activating predictive hypoglycemia shutdown (SAP-AAH)
  Interventions: Other: Brain MRI
- Control group (Other): age-matched control subjects without T1DM
  Interventions: Other: Brain MRI

INTERVENTIONS:
Device: AIDS — mylife CamAPS application, marketed by CamDiab Ltd, in conjunction with YpsoPump, marketed by Ypsomed, Dexcom blood glucose sensor, Orbit Infusion sets and Orbit Infusion sets and Orbit inserter (used in their indications)
  Other Names: Brain MRI
  Arms: AIDS group
Other: Brain MRI — To evaluate the neuroanatomical damage to gray matter associated with type 1 diabetes in young children according to their glycemic profile (AIDS use or not) and compared with an age-matched control subject

SUMMARY:
More than half of all new cases of type 1 diabetes (T1D) are diagnosed in the first decade of life. It has been reported that early onset T1D may be associated with deterioration in cognitive performance. It mainly affects working memory or the ability to perform complex tasks involving planning (executive functions) or decision-making. Brain magnetic resonance imaging (MRI) has reported alteration brain growth alteration related to impaired cognitive performance. Exposure to hypoglycemia, hyperglycemia and glycemic variability are thought to be responsible for these structural changes, especially in younger patients. Those changes can be detected early after diagnosis. Automatized insulin delivery systems (AIDS) can dramatically improve glycemic profile in children with T1D by reducing the occurrence of hypo and hyperglycemia. However, in France, market authorization are limited to children with unbalanced T1D who have failed to respond to other therapies and to the reinforcement of diabetes education. It therefore does not concern newly diagnosed patients. 60% of patients under 10 diagnosed with T1DM for less than 3 years are not treated in France by these systems. The aim of this study is therefore to determine whether early treatment of patients with AIDS would have a positive impact on cerebral growth and and on cognitive function in pediatric patients with T1DM.

DETAILED DESCRIPTION:
The aim of the study was to evaluate the neuroanatomical damage to gray matter associated with type 1 diabetes in young children according to their glycemic profile (use of a AIDS or Insulin pump combined with a continuous glucose monitoring sensor with the option of activating predictive shut-off before hypoglycemia (SAP-AAH)) and compared with an age-matched control subject.

Prospective case-control cohort study (T1DM or not) and exposed/non-exposed (CL or not), multicenter with 2 visits at 6 and 24 months of T1DM and 2 parallel visits for the control group.

The AIDS system used is a "mylife CamAPS application", marketed by CamDiab Ltd. class III, (YpsoPump, marketed by Ypsomed, Dexcom blood glucose sensor, used in their respective indications).

The experimental group will consist of patients treated with AIDS. The standard treatment (comparative) group will consist of patients with T1D treated with the gold standard treatment for this age group (SAP-AAH = insulin pump combined with a continuous glucose monitoring sensor with the option of activating predictive shut-off before hypoglycemia). In order to have a reference image, a second control group consisting of children aged 5 to 7 The expected benefits are early access to an automated insulin delivery system for study participants, as well as evidence of the neurocognitive benefit of early use of AIDs leading to changes in care practices.

ELIGIBILITY:
Inclusion Criteria:

* 5 to 7 years old
* Informed consent of parental guardians
* Parents able to speak, understand and read French (verified by investigator)
* Social security affiliation
* Only for subjects with T1DM:

  * Insulin pump treatment and Dexcom sensor wear
  * Type 1 diabetes diagnosed less than 6 months ago
  * Insulin dose ≥ 0.5 IU/k/day
  * Patients agree to use the DEXCOM sensor

Exclusion Criteria:

* History of neurological disease
* History of child psychiatric disease
* Prematurity (birth before 37 SA)
* Wearing of internal metal parts contraindicating the performance of MRI
* Severe skin disease preventing the use of an insulin pump sensor or catheter
* Uncontrolled celiac disease
* Uncontrolled autoimmune thyroiditis
* Participation in another interventional research study or in the exclusion period thereof
* Refusal to participate by a minor after information adapted to his/her age and abilities

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2028-03-20 (Estimated); Study Completion 2028-03-20 (Estimated)

PRIMARY OUTCOMES:
volume of total gray matter measured with high-resolution morphometric MRI | at inclusion and at 18 months after inclusion
  The primary endpoint will be changes in total gray matter volume measured with high-resolution morphometric MRI (vox based morphometry method).
  It will be measured at randomization (within 6 months of diagnosis) and 18 months after randomization in the intervention group (treatment of T1DM with SADI), in a control group of T1DM patients (treatment of T1DM with insulin pump and blood glucose sensor) and in a group of non-diabetic control subjects in the same age range.

SECONDARY OUTCOMES:
volume of total gray matter measured with high-resolution morphometric MRI | at month 6 and 24 months after diagnosis of T1DM
  Variation in other morphometric measures (localized gray matter, total and localized white matter, measurement of anatomical connectivity) and resting brain function (measurement of cerebral blood flow by arterial label spin ALS) will be compared between the two groups of diabetic children between randomization and the end of the 18-month intervention
Intelligence score | at month 6 and 24 months after diagnosis of T1DM
  Assessment of neurocognitive performance: Scale scores Wechsler Intelligence Scale for Children (WIPPSI-IV)
glycemic variability indexes | at month 6 and 24 months after diagnosis of T1DM
  Glycemic variability measured from data from continuous measurement of interstitial glycemia though the sensor worn by the patient. The standard deviation (SD) of the glycemic mean, the coefficient of variation (CV), the continuous overall net glycemic action (CONGA) 1 hour - 2 hours - 4 hours will be calculated from the full 72 hours recording closest to the visit. Their changes will be compared between the two measurement times between the groups.
Score of test "attention go/nogo" of KiTAP scale | at month 6 and 24 months after diagnosis of T1DM
  Behavioral control assessment and focused attention test
Score on BRIEF ((behavioral assessment inventory) scale | at month 6 and 24 months after diagnosis of T1DM
  behavioral assessment inventory
Score of Stroop big small et Stropp fruits scale | at month 6 and 24 months after diagnosis of T1DM
  Assessment of inhibitory control
Score of Nepsy II scale | at month 6 and 24 months after diagnosis of T1DM
  Auditory attention test

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Beltrand, PHD, Principal Investigator — APHP; Nathalie Boddaert, PHD, Study Chair — APHP
Locations (1):
- Hôpital Universitaire Necker Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No